CLINICAL TRIAL: NCT05918211
Title: Fontan Udenafil Exercise Longitudinal Assessment Trial (FUEL-2)
Brief Title: Fontan Udenafil Exercise Longitudinal Assessment Trial - 2
Acronym: FUEL-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mezzion Pharma Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MZ_Udenafil-05
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Single Ventricle Heart Disease
Keywords: Fontan; Maximal Oxygen Consumption; Work Rate; VO2 at VAT; Ventilatory Efficiency
MeSH Terms: interventions — udenafil

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled safety and efficacy study of udenafil versus placebo of approximately 436 subjects enrolled equally between the two arms (udenafil and placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active and matching placebo tablets will be identical in appearance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug (Experimental): Approximately 218 subjects dosed with udenafil will be enrolled at approximately 30 sites.
  Interventions: Drug: Udenafil
- Placebo (Experimental): Approximately 218 subjects dosed with matching placebo will be enrolled at approximately 30 sites.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Udenafil — Active drug
  Arms: Drug
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the clinical efficacy and safety of udenafil, an orally administered, potent and selective inhibitor of PDE5, versus placebo for the treatment of adolescent who have had the Fontan procedure.

DETAILED DESCRIPTION:
This study is a 26 week, prospective, multicenter, randomized, double-blinded, placebo-controlled safety and efficacy study of udenafil vs. placebo in adolescent subjects who have had the Fontan procedure. The primary efficacy endpoint will be change from baseline at 26 weeks in peak minute oxygen consumption (VO2 mL/kg/min) as measured by maximal cardiopulmonary exercise test (CPET) reading laboratory who will be blinded to treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females with Fontan physiology who are 12 to less than 19 years of age at enrollment.
2. Participant consent or parental/guardian consent and participant assent.
3. Participant fluency in primary language of country in which study is being conducted.
4. Current antiplatelet or anticoagulant therapy.

Exclusion Criteria:

1. Height < 132 cm.
2. Weight < 40 kg.
3. Hospitalization for acute decompensated heart failure within the last 12 months.
4. Current intravenous inotropic drugs.
5. Undergoing evaluation for heart transplantation or listed for transplantation.
6. Diagnosis of active protein losing enteropathy or plastic bronchitis within the last 3 years, or a history of liver cirrhosis.
7. Known Fontan baffle obstruction, branch pulmonary artery stenosis, or pulmonary vein stenosis resulting in a mean gradient of > 4 mmHg between the regions proximal and distal to the obstruction as measured by either catheterization or echocardiography, obtained prior to screening for the trial.
8. Single lung physiology with greater than 80% flow to one lung.
9. Failure to achieve maximal exertion (defined as RER < 1.10) on screening/baseline exercise test.
10. Peak minute oxygen consumption (VO2) less than 45% or ≥ 80% of predicated for age and gender at enrollment.
11. Severe ventricular dysfunction assessed qualitatively by clinical echocardiography within 6 months prior to enrollment.
12. Severe valvar regurgitation, ventricular outflow obstruction, or severe aortic arch obstruction assessed by clinical echocardiography within six months prior to enrollment.
13. History of significant renal (serum creatinine > 2.0), hepatic (serum AST and/or ALT > 3 times upper limit of normal), gastrointestinal or biliary disorders that could impair absorption, metabolism or excretion of orally administered medications.
14. Inability to complete exercise testing at baseline screening.
15. Subjects with a pacemaker whose heart rate at peak exercise is controlled by the extrinsic pacemaker as opposed to a native atrial rhythm.
16. History of PDE-5 inhibitor use within 12 months prior to enrollment. (Treatment is defined as chronic therapy as opposed to a single dose.)
17. History of any other medication for treatment of pulmonary hypertension within 3 months before study onset.
18. Known intolerance to oral udenafil.
19. Frequent use of medications or other substances that inhibit or induce CYP3A4.
20. Current use of alpha-blockers or nitrates.
21. Ongoing or planned participation in another research protocol that would either prevent successful completion of planned study testing or invalidate its results.
22. Noncardiac medical, psychiatric, and/or social disorder that would prevent successful completion of planned study testing or would invalidate its results.
23. Cardiac care, ongoing or planned, at a non-study center that would impede study completion.
24. For females: Pregnancy at the time of screening, pregnancy planned before study completion, or refusal to use an acceptable method of contraception for study duration if sexually active.
25. Unable to abstain or limit intake of grapefruit juice and grapefruit containing drinks during the duration of the trial.
26. Refusal to provide written informed consent/assent.
27. In the opinion of the investigator, the subject is likely to be non-compliant with the study protocol.
28. History of clinically significant thromboembolic event, in the option of the site Principal Investigator, that may put the subject at increased risk of a subsequent event while participating in the study.
29. Coronavirus disease 2019 (COVID-19) vaccination or symptoms of COVID-19 infection within 7 days of Visit 1.
30. Not taking antiplatelet or anticoagulant therapy.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 436 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-10-28 (Estimated); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
Change in Exercise Capacity | Baseline to 26 Weeks
  The change in exercise capacity (as measured by maximal VO2 at maximum exercise effort) from baseline to 26 weeks (or study completion)

SECONDARY OUTCOMES:
Change in VO2 at the ventilatory anaerobic threshold (VAT) | Baseline to 26 weeks
  Change in peak oxygen consumption (VO2) from baseline to Week 26 as measured by maximal central cardiopulmonary exercise test (CPET) reading laboratory.
Change in Enhanced Liver Fibrosis (ELF) Score | Baseline to 26 weeks
  Change from baseline to Week 26 in the Enhanced Liver Fibrosis (ELF) Score calculated by the change in the following biomarkers: hyaluronic acid, amino-terminal propeptide of type III collagen, and tissue inhibitor of metalloproteinase-1. subjects with scores of <7.7 were assigned to the no or mild fibrosis group; 7.7 to 9.8 to the moderate fibrosis group, and >9.8 to the severe fibrosis group.
Work rate (watts) at ventilatory anaerobic threshold (VAT) | Baseline to 26 weeks
  Change from baseline to 26 weeks in work rate in watts at the ventilatory anaerobic threshold as measured by the central cardiopulmonary exercise test reading laboratory.
Change in ventilatory efficiency (VE/VCO2) at ventilatory anaerobic threshold | Baseline to 26 weeks
  Change from baseline to Week 26 in ventilatory efficiency calculated by ventilatory efficiency divided by minute carbon dioxide production at the ventilatory anaerobic threshold (VE/VCO2 at VAT).

CONTACTS AND LOCATIONS:
Overall Officials: WG Kim, Study Director — Mezzion Pharma Co. Ltd
Locations (40):
- United States (37):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital of Colorado, Denver, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Nemours Children's Hospital, Wilmington, Delaware
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - UF Health Shands Hospital, Gainesville, Florida
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Hospital of Georgia, Augusta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Mercy Hospital Kansas City, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska Children's Hospital and Medical Center, Omaha, Nebraska
  - Mt. Sinai Children's Hospital, New York, New York
  - New York-Presbyterian Children's Hospital, New York, New York
  - Dana.Amaro@atriumhealth.org, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - MUSC Pediatric Research Group, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- South Korea (3):
  - Sejong General Hospital, Bucheon-si, Gyeonggi-do
  - Seoul National University Children's Hospital, Seoul
  - Yonsei Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No